CLINICAL TRIAL: NCT04698382
Title: Impact of COVID-19 on the Incidence, Characteristics, Management and Outcome of Sepsis
Status: Withdrawn | Type: Observational
Why Stopped: Reduced relevance due to end of pandemic
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Sameer Kadri, M.D., Staff Clinician, Critical Care Medicine Department, National Institutes of Health Clinical Center (CC)
Other Study IDs: BD022384
Record Dates: First submitted 2021-01-05; First posted 2021-01-06 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Sepsis; Septic Shock
Keywords: sepsis; septic shock; COVID-19
MeSH Terms: conditions — Sepsis; Shock, Septic; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-COVID-19-related sepsis: Non-COVID-19 sepsis patients will be identified with sepsis or septic shock without a COVID-19 diagnosis code or a positive COVID-19 laboratory test.
  Sepsis patients will be defined as patients with concurrent infection and organ dysfunction. Presumed concurrent infection will be defined as a blood culture order and ≥ 3 days of antibiotics administration, including at least 24h of intravenous antibiotics, or death while on antibiotics within 3 days of admission. Organ dysfunction will be defined by ICD-10-modified acute organ failure score. Sensitivity analyses will use ICD-10 explicit sepsis codes to define non-COVID-19 sepsis instead.
  COVID-19 will be identified based on receiving a diagnosis code for COVID-19 (U07.1) or legacy coding (prior to the implementation of a specific COVID-19 code) present-on-admission and/or a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) polymerase chain reaction (PCR) test on admission
- Non-COVID-19, Non-Sepsis Control Population: This will be defined as patients identified with emergency conditions of interest without a diagnosis code of sepsis, COVID19 or a positive COVID-19 laboratory test.
  These include
  1. Acute Gastrointestinal Bleeding (GIB): Patients with at least one GIB ICD-10 code and one relevant CPT intervention codes.
  2. Myocardial Infarction (MI): Patients with at least one MI ICD-10 code and one relevant CPT intervention codes

SUMMARY:
This study seeks to determine the the impact of COVID-19 on the incidence, characteristics, management and outcome of patients admitted to U.S. hospitals with non-COVID-19 related sepsis.

DETAILED DESCRIPTION:
Sepsis is the most common cause of death and the most expensive condition among hospitalized patients in the U.S. The delivery of high-quality care for sepsis necessitates optimal institutional functionality and availability of adequate healthcare personnel and resources. However, since the novel coronavirus disease 2019 (COVID-19) pandemic hit the U.S., fear of acquisition of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has resulted in fewer patients with acute conditions seeking hospitalization. Furthermore, the rapid onslaught of COVID-19 admissions has profoundly strained hospital supplies, personnel and care processes and left little time to re-calibrate the management of other acute conditions that share these resources. As such, the impact on the detection, triage, monitoring, resuscitation, and outcome of patients with sepsis is currently unknown. Large administrative and clinical data repositories of inpatient discharges that are populated in near-real time may enable study of contemporaneous inpatients with COVID-19 and sepsis (without COVID-19) respectively.

We aim to:

Aim 1: Determine the impact of the COVID-19 pandemic on the incidence of hospital admission for non-COVID-19-related sepsis and septic shock and the proportion of these patients that receive Intensive Care Unit-level care. This analysis will assess for dynamic changes in the number of patients developing and/or seeking hospital care for sepsis and septic shock during the pandemic and whether the burden of critically ill and mechanically ventilated patients with COVID-19 may have impacted the threshold for providing ICU-level care to patients with sepsis and septic shock

Aim 2: Determine the trend in risk-adjusted mortality among patients admitted with non-COVID-19-related sepsis and septic shock during the pandemic. This analysis will indicate whether being hospitalized for sepsis/septic shock during vs. prior to the pandemic was associated with any change survival. An analysis will be performed to identify prognostic factors associated with non-COVID-19-related sepsis and septic shock.

Aim 3: Determine the impact of COVID-19-specific center-level characteristics (e.g. case volume, multi-ICU status, intubation threshold) on risk-adjusted mortality of non-COVID-19-related sepsis and septic shock during the pandemic period. Identification and modification of pandemic-related triage and processes that impact survival in sepsis may help preserve quality of care when health systems are strained.

Aim 4: Determine the impact of COVID-19 on processes of care in the management of sepsis: This aim will investigate whether COVID-19 has impacted key quality processes in the management of patients with sepsis present on admission (POA).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to U.S hospitals with sepsis (without COVID-19)
* Patients admitted to U.S hospitals with acute gastrointestinal bleeding (without COVID-19 or sepsis)
* Patients admitted to U.S hospitals with sepsis myocardial infarction (without COVID-19 or sepsis)

Exclusion Criteria:

* Patients admitted to U.S. hospitals with COVID-19
* Patients with acute gastrointestinal bleeding with sepsis or COVID-19
* Patients with myocardial infarction with sepsis or COVID-19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Non-COVID-19-related sepsis This will be defined as patients identified with sepsis or septic shock without a diagnosis code of COVID-19 or a positive COVID-19 laboratory test.
  Non-COVID-19, Non-Sepsis Control Population This will be defined as patients identified with emergency conditions of interest without a diagnosis code of sepsis, COVID19 or a positive COVID-19 laboratory test.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of hospital and ICU Admission | From admission to in-hospital death or discharge to hospice
  Determine the impact of the COVID-19 pandemic on the incidence of hospital admission for non-COVID-19-related sepsis and septic shock and the proportion of these patients that receive Intensive Care Unit-level care
In-hospital Mortality | From admission to in-hospital death or discharge to hospice
  Determine the trend in risk-adjusted in-hospital mortality (or discharge to hospice) among patients admitted with non-COVID-19-related sepsis and septic shock

SECONDARY OUTCOMES:
Sepsis management quality metrics | From time of admission to death during the hospitalization
  Determine the impact of COVID-19 on quality metrics in the management of sepsis patients

CONTACTS AND LOCATIONS:
Overall Officials: Sameer S Kadri, MD, MS, Principal Investigator — National Institutes of Health, Clinical
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
N/A this data is deidentifed